CLINICAL TRIAL: NCT00267787
Title: Molecular Genetic and Pathological Studies of Anal Tumors
Status: Terminated | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: ANAL0001; 95340 (Other: Stanford University Alternate IRB Approval Number); ANAL0001 (Other: Stanford University); 14037 (Other: Stanford IRB)
Record Dates: First submitted 2005-12-19; First posted 2005-12-21 (Estimated); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Rectal Cancer; Colon Cancer; Colonic Neoplasms; Anal Cancer
MeSH Terms: conditions — Rectal Neoplasms; Colonic Neoplasms; Anus Neoplasms | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: genetic analysis — standard of care

SUMMARY:
Study the Genetics of Anal Cancer

DETAILED DESCRIPTION:
To determine the status of previously identified anal cancer molecular markers and any correlations with outcome as well as to discover new molecular biomarkers through correlating molecular data with clinical outcome. Study of tissue samples and cells from biopsies of your lesion and blood sample. We hope to learn the role genes and proteins may play in the development of anal cancer. Experiments will be performed using this tissue and blood, include analysis of DNA, analysis of RNA expression levels, analysis of protein levels of important gene products, and development of tissue culture cell lines.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria:

* Patients with anal tumors
* Undergoing surgery for elective colon and rectal surgery Exclusion Criteria:No other patients other than adult patients with anal cancer or high risk for anal cancer refered to Stanford will be enrolled to the study. No Children will be included to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with anal cancer or high risk for anal cancer refered to Stanford.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2004-09; Primary Completion 2012-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Genetic analysis of blood sample as well as tissues , will provide us with any possible tumor marker for a better prognostic indicator. | Annual assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lane Welton, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No